CLINICAL TRIAL: NCT02544438
Title: a Phase i/Iia, Open Label, Uncontrolled Study to Evaluate the Safety and Efficacy of Astarabine (BST-236) as Single Agent in Patients With Refractory or Relapsed Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL) Disease
Brief Title: Study Evaluating the Safety and Efficacy of Astarabine in Acute Myeloid Leukemia or Acute Lymphoblastic Leukemia
Acronym: BSTPHASE1-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioSight Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BST-PHASE1-01
Record Dates: First submitted 2015-08-23; First posted 2015-09-09 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Astarabine (Experimental): Astarabine
  Interventions: Drug: Astarabine (BST-236)

INTERVENTIONS:
Drug: Astarabine (BST-236) — Cohort # Astarabine Dose Number of Patients
  1. 0.5 gr/m2 (0.3 age>50) 3
  2. 1.5 gr/m2(0.8age>50) 3
  3. 3.0 gr/m2(1.5 age>50) 3
  4. 4.5 gr/m2(2.3 age>50) 6
  5. 4.5 gr/m2 (no age limit) 3 up to 6
  6. 6 gr/m2 (no age limit) 3 up to 6
  Total number of patients: up to 24

SUMMARY:
A Phase I/IIa, open-label, uncontrolled study to evaluate the safety and efficacy of Astarabine (BST-236) as single agent in patients with refractory or relapsed Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL) disease

DETAILED DESCRIPTION:
This is prospective, Phase I/IIa, open-label, uncontrolled, single-center, single arm study to evaluate the safety and efficacy of Astarabine given intravenously (I.V.) in escalated doses for 6 days for cycle in patients with relapsed or refractory AML or ALL who are more than 18 years of age. Patients will be screened for eligibility based on existing records and/or specific laboratory examinations performed for the screening process.

Patients will be gradually enrolled into 4 subsequent cohorts of escalating drug doses:

Cohort # Astarabine Dose Number of Patients

1. 0.5 gr/m2 (0.3 age>50) 3
2. 1.5 gr/m2 (0.8age>50) 3
3. 3.0 gr/m2 (1.5 age>50) 3
4. 4.5 gr/m2 (2.3 age>50) 6
5. 4.5 gr/m2 (no age limit) 3 up to 6
6. 6 gr/m2 (no age limit) 3 up to 6

Maximal tolerated dose (MTD) will be defined in case 2 subjects will experience a dose limiting toxicity (DLT)

ELIGIBILITY:
Inclusion Criteria:

1. A. Relapsed or refractory acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL), based on World Health Organization Classification; Patients must have morphological proof of AML or ALL with blasts in peripheral blood (PB) or 5% in bone marrow (BM) within 2 weeks prior to study registration.

   I. Refractory disease will be considered failure to either respond to induction chemotherapy and/or salvage therapy.

   II. 2nd relapse III. Relapse following autologous or allogeneic stem cell transplantation. B. patients which at the physician discretion are not eligible for standard chemotherapy, whether induction or consolidation, due to age or significant co-morbidities
2. Age ≥18 years.
3. Ability to understand and willingness to sign the written informed consent document.
4. Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment and use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
5. Male subject agrees to use an acceptable method for contraception for the duration of the study.
6. Eastern cooperative oncology group (ECOG) performance status ≤ 2
7. Hydroxyurea is permitted to control high white blood cells (WBC) count prior to study entry.
8. Previous treatment related toxicities must have resolved to less than Grade 2 (excluding alopecia).

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. l. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, uncontrolled hypertension, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
2. Patients with compromised pulmonary function who needs oxygen therapy.
3. Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
4. Patients who have had chemotherapy (except for hydroxyurea), biologic therapy, immunotherapy, or radiotherapy within 2 weeks of induction therapy or 4 weeks of consolidation or intensive therapy (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
5. Patients receiving any other investigational agents.
6. Patients who have had any surgical procedure, excluding central venous catheter placement or other minor procedures (e.g. skin biopsy) within 14 days of Day 1.
7. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
8. Patients with prior malignancy are eligible; however, the patient must be in remission from the prior malignancy and have completed all chemotherapy and radiotherapy at least 6 months prior to registration and all treatment-related toxicities must have resolved.
9. Leptomeningeal/ central nervous system involvement with AML; a lumbar puncture does not need to be performed unless there is clinical suspicion.
10. Patients with active central nervous system disease or with granulocytic sarcoma as sole site of disease.
11. Patients who have had prior pulmonary radiation.
12. Liver enzymes (AST and alanine aminotransferase (ALT) more than 2.5 times the upper limits of normal (ULN), and total bilirubin more than 1.5 x ULN within 14 days of enrollment.
13. Renal function: Serum creatinine more than 1.5 x ULN within 24 hours of enrollment.
14. Existence of inter-current organ damage or medical condition that would prohibit or interfere with study drug therapy.
15. If the patient has co-morbid medical illness, life expectancy attributed to this must be greater than 3 months.
16. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Astarabine/Ara-C.
17. Pregnant women are excluded from this study because Astarabine/Ara-C are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Astarabine, breastfeeding should be discontinued if the mother is treated with Astarabine.
18. known history of Human immunodeficiency virus (HIV) or active hepatitis B or C
19. Concurrent use of the following medications: Digoxin, Gentamycin, fluorocytosine, L-asparginase, any drugs or supplements that interfere with blood clotting can raise the risk of bleeding during treatment with Ara-C. These include: vitamin E, non-steroidal anti-inflammatory drugs (NSAIDs) such as aspirin, warfarin, ticlopidine, clopidogrel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) | 90 days
Dose limiting Toxicity (DLTs) | within 90 days
  Any ≥ grade 3 non-hematologic toxicity (excluding alopecia, hypersensitivity) Grade 3 nausea and vomiting if it occurs despite maximal (5HT antagonist and corticosteroid) antiemetic therapy, and if hydration is required for >24 hours.
  Grade 3 diarrhea despite patient compliance with loperamide therapy.

SECONDARY OUTCOMES:
safety and tolerability expressed by any grade adverse events (AEs) | within 90 days
PharmacoKintetics (PK): maximum plasma concentration (Cmax) | PK studies will be performed up to 8 days at the following time points: 0', 15', 30', 60', 90', 120', 240', 360', and 600' of days: 1 to 6 and 24 hours and 48 hours after last Astarabine administration (days 7 - 8)
response rate: complete remission + partial remission (CR + PR) | within 90 days
  using the revised recommendations of the international working group for diagnosis, standardization of response criteria, tratment outcome and reporting stanndadarts fro therapeutic trials in acute myeloid leukemia
Phrmacokinetics (PK): area under the curve (AUC) versus time curve | PK studies will be performed up to 8 days at the following time points: 0', 15', 30', 60', 90', 120', 240', 360', and 600' of days: 1 to 6 and 24 hours and 48 hours after last Astarabine administration (days 7 - 8)

CONTACTS AND LOCATIONS:
Overall Officials: Tsila Zuckerman, MD, Principal Investigator — Rambam Health Care Campus
Locations (2):
- Israel (2):
  - Rambam medical center hematology department, Haifa
  - Tel Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Derived] Zuckerman T, Ram R, Akria L, Koren-Michowitz M, Hoffman R, Henig I, Lavi N, Ofran Y, Horowitz NA, Nudelman O, Tavor S, Yeganeh S, Gengrinovitch S, Flaishon L, Tessler S, Ben Yakar R, Rowe JM. BST-236, a novel cytarabine prodrug for patients with acute leukemia unfit for standard induction: a phase 1/2a study. Blood Adv. 2019 Nov 26;3(22):3740-3749. doi: 10.1182/bloodadvances.2019000468. PMID 31770437